CLINICAL TRIAL: NCT04895904
Title: Endoscopic Diagnosis, Treatment and Prognosis of Acute Nonvariceal Upper Gastrointestinal Bleeding in Nanchang, Jiangxi Province, China.
Brief Title: Endoscopic Diagnosis and Treatment of Acute Nonvariceal Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xu Shu, Professor, The First Affiliated Hospital of Nanchang University
Other Study IDs: 2021058
Record Dates: First submitted 2021-05-19; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Acute Upper Gastrointestinal Non Variceal Hemorrhage
Keywords: Acute upper gastrointestinal non variceal hemorrhage; peptic ulcer; Dieulafoy's lesion; Gastric ulcer bleeding; Endoscopic hemostasis
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Our study is an observational study and the main purpose of our study is to observe the efficacy of endoscopic hemostasis and drug therapy

SUMMARY:
Acute nonvariceal upper gastrointestinal bleeding (ANVUGIB) is a common critical disease in gastroenterology. Due to the development of modern medical technology, the incidence rate of ANVUGIB has been decreasing in recent years, but its mortality within 30 days is still 11%. Endoscopic hemostasis and drug therapy are the first choice for the treatment of ANVUGIB. After endoscopic hemostasis, it is very important to treat peptic ulcer bleeding with strong acid suppression therapy to maintain gastric pH above 6.0. This study is to study the effect of endoscopic and drug treatment of ANVUGIB.

DETAILED DESCRIPTION:
Acute nonvariceal upper gastrointestinal bleeding (ANVUGIB) is a common critical disease in gastroenterology. It refers to the bleeding caused by the non varicose diseases above the ligament of flexor, including the bleeding of pancreaticobiliary tract and the bleeding caused by the diseases near the anastomotic stoma after gastrojejunostomy. Due to the development of modern medical technology, the incidence rate of ANVUGIB has been decreasing in recent years. A US study shows that the incidence rate of ANVUGIB dropped from 78/10 to 61/10 10000 [1] from 2001 to 2009. However, the mortality within 30 days of ANVUGIB is still as high as 11% [2]. Peptic ulcer bleeding is the most common cause of bleeding in ANVUGIB. The annual incidence rate is 19.4-57/10 million, and the rate of rebleeding within 7 days is 13.9%, and the mortality rate is 30 in 30 days. A study in China shows that compared with the 1990s, the detection rate of high-risk ulcer has increased, but the overall mortality has not decreased significantly [4]. Endoscopic hemostasis is the first choice for the treatment of peptic ulcer. The latest guidelines of our country recommend that patients with upper gastrointestinal bleeding with stable hemodynamics should try their best to have emergency gastroscopy within 24 hours after bleeding, and emergency endoscopic hemostasis is feasible for bleeding lesions [5]. After endoscopic hemostasis, it is very important to give strong acid suppression therapy to maintain gastric pH above 6.0 in the treatment of peptic ulcer bleeding [6-9]. This study is to analyze the effect of endoscopic and drug treatment of ANVUGIB.

ELIGIBILITY:
Inclusion Criteria:

* From January 2014 to February 2021, patients with acute nonvariceal upper gastrointestinal bleeding underwent emergency endoscopic hemostasis in our hospital.

Exclusion Criteria:

* 1. The age is less than or equal to 18 years old and greater than or equal to 85 years old; 2. Forrest grade IIC and III; 3. Complicated with severe cardiovascular and cerebrovascular diseases or severe liver and kidney diseases (such as heart failure, liver failure, renal failure, etc.); 4. The records of the cases were incomplete.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The people who come to Nanchang University First Affiliated Hospital for medical treatment
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Rebleeding | Within 30 days after endoscopic hemostasis
  Clinically, the following symptoms or laboratory examination results suggest rebleeding within 30 days after successful endoscopic hemostasis：(1) The frequency of hematemesis or melena increased, the vomit was bright red or dark red bloody stool, or accompanied by active bowel sounds;
  (2) After rapid infusion and blood transfusion, the symptoms of peripheral circulation failure did not improve significantly, or although temporarily improved and then deteriorated, the central venous pressure still fluctuated, slightly stable and then decreased;
  (3) Red blood cell count, hemoglobin concentration and hematocrit continued to decrease, reticulocyte count continued to increase;
  (4) In the case of sufficient fluid replacement and urine volume, blood urea nitrogen continued or increased again.

SECONDARY OUTCOMES:
surgery due to rebleeding | Within 30 days after endoscopic hemostasis
  Surgical treatment for rebleeding
Mortality | Within 30 days after endoscopic hemostasis
  Mortality due to rebleeding

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to make it public. Please contact me if you need

REFERENCES:
- [Result] Laine L, Yang H, Chang SC, Datto C. Trends for incidence of hospitalization and death due to GI complications in the United States from 2001 to 2009. Am J Gastroenterol. 2012 Aug;107(8):1190-5; quiz 1196. doi: 10.1038/ajg.2012.168. Epub 2012 Jun 12. PMID 22688850
- [Result] Rosenstock SJ, Moller MH, Larsson H, Johnsen SP, Madsen AH, Bendix J, Adamsen S, Jensen AG, Zimmermann-Nielsen E, Nielsen AS, Kallehave F, Oxholm D, Skarbye M, Jolving LR, Jorgensen HS, Schaffalitzky de Muckadell OB, Thomsen RW. Improving quality of care in peptic ulcer bleeding: nationwide cohort study of 13,498 consecutive patients in the Danish Clinical Register of Emergency Surgery. Am J Gastroenterol. 2013 Sep;108(9):1449-57. doi: 10.1038/ajg.2013.162. Epub 2013 Jun 4. PMID 23732464
- [Result] Barkun AN, Almadi M, Kuipers EJ, Laine L, Sung J, Tse F, Leontiadis GI, Abraham NS, Calvet X, Chan FKL, Douketis J, Enns R, Gralnek IM, Jairath V, Jensen D, Lau J, Lip GYH, Loffroy R, Maluf-Filho F, Meltzer AC, Reddy N, Saltzman JR, Marshall JK, Bardou M. Management of Nonvariceal Upper Gastrointestinal Bleeding: Guideline Recommendations From the International Consensus Group. Ann Intern Med. 2019 Dec 3;171(11):805-822. doi: 10.7326/M19-1795. Epub 2019 Oct 22. PMID 31634917
- [Result] Lanas A, Dumonceau JM, Hunt RH, Fujishiro M, Scheiman JM, Gralnek IM, Campbell HE, Rostom A, Villanueva C, Sung JJY. Non-variceal upper gastrointestinal bleeding. Nat Rev Dis Primers. 2018 Apr 19;4:18020. doi: 10.1038/nrdp.2018.20. PMID 29671413
- [Result] Canamares-Orbis P, Chan FKL. Endoscopic management of nonvariceal upper gastrointestinal bleeding. Best Pract Res Clin Gastroenterol. 2019 Oct-Dec;42-43:101608. doi: 10.1016/j.bpg.2019.04.001. Epub 2019 Apr 17. PMID 31785733
- [Derived] Lai Y, Xu Y, Zhu Z, Pan X, Long S, Liao W, Li B, Zhu Y, Chen Y, Shu X. Development and validation of a model to predict rebleeding within three days after endoscopic hemostasis for high-risk peptic ulcer bleeding. BMC Gastroenterol. 2022 Feb 14;22(1):64. doi: 10.1186/s12876-022-02145-9. PMID 35164682